CLINICAL TRIAL: NCT06747676
Title: Graviceptive Neglect After Stroke: Clinical, Neuroanatomical and Physiological Effects of Focal Neuromodulation
Brief Title: GRAViceptive NEGlect Treatment in Acute Stroke Using Targeted Cranial ELECTrotherapy
Acronym: GravNegElect
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Thomas Jefferson University (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Viasonix (Unknown); Phelcom (Unknown); FBX Medical (Unknown)
Responsible Party: Principal Investigator, Taiza G. S. Edwards, PhD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 74877723.4.0000.5440; 2023/03252-2 (Other Grant/Funding Number: The São Paulo Research Foundation)
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Stroke
Keywords: Stroke; Graviceptive Neglect; Verticality Perception; Non-invasive Brain Stimulation; Neuroimaging; Electroencephalography; Transcranial doppler; HD-tDCS
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Phase I/II randomized sham-controlled double-blind parallel clinical trial design
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active HD-tDCS (Experimental): Participants will receive six sessions of 2mA active HD-tDCS cathode center over the contralesional TPJ for 20 minutes, 3 times daily for 2 days with session intervals greater than 3 hours.
  Interventions: Device: Active: High-Definition transcranial Direct Current Stimulation (HD-tDCS)
- Sham HD-tDCS (Sham Comparator): Participants will receive six sessions of 2mA sham HD-tDCS cathode center over the contralesional TPJ for 20 minutes, 3 times daily for 2 days with session intervals greater than 3 hours.
  Interventions: Device: Sham: High-Definition transcranial Direct Current Stimulation (HD-tDCS)

INTERVENTIONS:
Device: Active: High-Definition transcranial Direct Current Stimulation (HD-tDCS) — Active high-definition transcranial direct current stimulation (HD-tDCS) will be delivered by a low-intensity direct current stimulator (Soterix Medical) using a 3x1 ring configuration with a central cathode over the contralesional temporo-parietal junction. During the stimulation, participants will perform tasks to stimulate correct visual verticality perception. Six active HD-tDCS sessions of 2mA for 20 minutes HD-tDCS, 3 times daily for 2 days with session intervals greater than 3 hours.
  Arms: Active HD-tDCS
Device: Sham: High-Definition transcranial Direct Current Stimulation (HD-tDCS) — Six sessions (3 times daily for 2 days) of 2mA sham HD-tDCS cathode center over the contralesional TPJ for 20min. Direct current (DC) will be generated by a low-intensity direct current stimulator (Soterix Medical) and then split into the 3 high-density Ag/AgCl sintered ring electrodes. The sham stimulation condition will consist of the same positioning of the electrodes as the active condition, with a ramp-up to 2mA over 30 seconds and a subsequent ramp-down of 30 seconds.
  Arms: Sham HD-tDCS

SUMMARY:
We aim to determine if targeted high-definition transcranial direct current stimulation (HD-tDCS) can safely correct errors in visual verticality perception in patients after stroke affecting either hemisphere.

DETAILED DESCRIPTION:
This study explores a new approach to treat graviceptive neglect, a condition that affects balance and perception of uprightness, using a non-invasive brain stimulation technique called HD-tDCS (high-definition transcranial direct current stimulation). Using a phase I/II randomized sham-controlled double-blind parallel clinical trial design, we aim to analyze if HD-tDCS can safely help correct abnormal visual verticality perception in 28 people after stroke. We will also investigate the effects of our protocol on cerebrovascular response using transcranial Doppler and cortical activity using EEG. Neuroanatomical characteristics will be analyzed to establish the relationship between verticality perception error and the extent of temporo-parietal junction (TPJ) damage and, more broadly, the putative VV structural brain Network (VVN). Each participant will receive six HD-tDCS sessions of 2mA for 20 minutes in a central cathode montage applied over the contralesional TPJ. Patients will be randomized into two groups, with 50% receiving active stimulation and 50% receiving sham stimulation. The sham stimulation condition will consist of the same electrode placement, with a 2mA ramp-up over 30 seconds, followed by a 30-second ramp-down. Both groups will undergo 6 sessions, three times a day, for 2 days. The follow-up assessment will be performed 1 month after stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Supratentorial ischemic stroke diagnosed by neuroimaging and clinical analysis;
* Clinically stable (stable vital signs for 24 hours; no chest pain in the last 24 hours; no significant arrhythmia; no evidence of deep vein thrombosis);
* Normal or corrected-to-normal vision;
* No previous experience with HD-tDCS;
* Ability to provide informed consent (patient or legal representative);
* Ability to comply with the intervention and assessment schedule of the protocol.
* Presence of visual verticality misperception.

Exclusion Criteria:

* Migraine;
* Pregnancy;
* Pacemakers;
* Seizures;
* Claustrophobia;
* Transient ischemic attack;
* Other neurological disorders;
* Psychiatric disorders;
* Sensitive scalp or prior brain surgery;
* Diagnosis of severe carotid atherosclerotic disease (stenosis ≥ 70%);
* Presence of metal implants, cardiac pacemakers, or claustrophobia;
* Diagnosis of COVID-19 or other infectious disease that requires isolation;
* Uncontrolled medical problems, such as terminal cancer or kidney disease.
* Left-handed or mixed-handed individuals as determined using the Edinburgh Handedness Inventory (Appendix 10);
* Peripheral vestibular deficits observed using neuro-otological screening tests when the participant's clinical condition allows (head shake test, head thrust test, Dix-Hallpike, and Pagnini-McClure);
* Prior musculoskeletal disorders affecting alignment and postural balance (e.g., moderate to severe scoliosis; torticollis);
* Cognitive dysfunction outside normal limits on the Mini-Mental State Examination (score below 23);
* Global or Wernicke's aphasia;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Visual Verticality Perception (VV; visual graviceptive neglect) | From baseline (before the first session) to 1 day post-intervention protocol (after six HDtDCS sessions).
  Change in VV: assessment using the bucket method.

SECONDARY OUTCOMES:
Visual Verticality Perception (VV; visual graviceptive neglect) | From baseline (before the first session) to 30±5 days post-intervention protocol (after six HDtDCS sessions).
  Change in VV: assessment using the bucket method.
Ocular torsion | From baseline (before the first session) to 1 day post-intervention protocol (after six HDtDCS sessions).
  Change in ocular torsion: assessment using fundus photography (Phelcom; Eyer 1 device)
Ocular torsion | From baseline (before the first session) to 30±5 days post-intervention protocol (after six HDtDCS sessions).
  Change in ocular torsion: assessment using fundus photography (Phelcom; Eyer 1 device)
Electroencephalography | From baseline (before the first session) to 1 day post-intervention protocol (after six HDtDCS sessions).
  Electroencephalography measurements focusing on resting state networks related to visual verticality perception.
Electroencephalography | From baseline (before the first session) to 30±5 days post-intervention protocol (after six HDtDCS sessions).
  Electroencephalography measurements focusing on resting state networks related to visual verticality perception.
Cerebrovascular reactivity | From baseline (before the first session) to 1 day post-intervention protocol (after six HDtDCS sessions).
  Transcranial Doppler Ultrasonography (TCD; Viasonix Dolphin/XF Robot) will be employed to measure cerebral blood flow velocity in the middle cerebral arteries while the participant performs the breath-holding maneuver.
Cerebrovascular reactivity | From baseline (before the first session) to 30±5 days post-intervention protocol (after six HDtDCS sessions).
  Transcranial Doppler Ultrasonography (TCD; Viasonix Dolphin/XF Robot) will be employed to measure cerebral blood flow velocity in the middle cerebral arteries while the participant performs the breath-holding maneuver.
Spatial neglect | From baseline (before the first session) to 1 day post-intervention protocol (after six HDtDCS sessions).
  Spatial neglect will be assessed using the conventional Behavior Inattention Test (BIT), which consists of 6 items: 1) line crossing; 2) letter cancellation; 3) star cancellation; 4) figure and shape copying; 5) line bisection; and 6) representational drawing.
Spatial neglect | From baseline (before the first session) to 30±5 days post-intervention protocol (after six HDtDCS sessions).
  Spatial neglect will be assessed using the conventional Behavior Inattention Test (BIT), which consists of 6 items: 1) line crossing; 2) letter cancellation; 3) star cancellation; 4) figure and shape copying; 5) line bisection; and 6) representational drawing.

OTHER OUTCOMES:
Brain magnetic resonance imaging (MRI) | Up to 15 days post stroke.
  The structural integrity of the visual verticality network will be evaluated using diffusion MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Taiza Edwards, PhD, Principal Investigator — Ribeirão Preto Medical School, University of São Paulo
Locations (2):
- Brazil (2):
  - Ribeirão Preto Medical School, University of São Paulo, Ribeirão Preto, São Paulo
  - University of São Paulo, Ribeirão Preto Medical School, Ribeirão Preto, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided